CLINICAL TRIAL: NCT04478851
Title: Project EXCEL: Dissemination, Implementation, and Effectiveness of the Exercise Oncology Survivorship Partnership Model - Reaching Rural Cancer Survivors to Enhance Quality of Life
Brief Title: EXCEL: Exercise for Cancer to Enhance Living Well
Acronym: EXCEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); Dalhousie University (Other); Alberta Health services (Other); University Health Network, Toronto (Other); Memorial University of Newfoundland (Other); University of British Columbia (Other); University of Prince Edward Island (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-20-0098
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Head and Neck Cancer; Colon Cancer; Breast Cancer; Prostate Cancer; Cancer Caregivers
Keywords: Physical activity; Exercise; Community programs; Online resources; Quality of life; Cancer survivor; mobile health; telehealth
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms; Colonic Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Hybrid implementation effectiveness study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will be involved in group exercise classes, twice a week for 12 weeks.
  Interventions: Behavioral: Group Exercise Classes

INTERVENTIONS:
Behavioral: Group Exercise Classes — The exercise program to be implemented for rural cancer survivors will combine aerobic, resistance, balance, and flexibility exercises delivered in a circuit-type class setting or group personal training format, twice weekly for a 12-week period. If public health restrictions require closure of fitness facilities due to COVID-19, the program will be delivered online. If facilities are open, the sessions will be integrated in the community, delivered in-person. Whether delivered in-class or remotely, the program follows exercise progression principles (ie, frequency, intensity, time, type, overload and progression) over the 12-weeks, with tailoring of any exercise to meet individual participant needs as required, in order to promote fitness and wellness benefits. The exercise intervention is based on the Alberta Cancer Exercise (ACE) program.

SUMMARY:
Project EXCEL will provide community or online exercise programs to rural and remote and under-served cancer survivors, as well as encourage participants to become life-long exercisers. Exercise is an evidence-based self-management strategy that benefits all cancer survivors. However, most cancer survivors who live in remote or rural places don't have adequate opportunities to be involved in exercise programs that are tailored to their needs.

DETAILED DESCRIPTION:
As cancer survivorship numbers grow, a focus on positive health in survivorship is essential. Exercise is an evidence-based effective self-management strategy that benefits all cancer survivors (CS). However, the majority of research and the limited development of evidence-based clinical or community programs in exercise and cancer has been conducted almost exclusively in urban academic and clinical settings, with very limited implementation outreach to "hard to reach" CS.

In this proposed cancer exercise hybrid implementation effectiveness research, over 5 years we will use an integrated knowledge translation approach to move the current evidence-base that clearly supports the role of exercise in cancer survivorship, into sustainable and effective community-based or online settings that will optimize the delivery of exercise to rural/remote and underserved CS (RCS). Implementing and evaluating the proposed Exercise Oncology Survivorship (EOS) partnership model will result in a sustainable resource to support the implementation and delivery of exercise oncology programs in rural Canadian communities.

Investigators will work to develop lasting referral pathways between cancer care clinics and local fitness professionals. These fitness professionals will have additional cancer specific training to ensure they can effectively and safely deliver the program. Eligible and consenting participants will be screened for exercise safety, and following fitness testing will be triaged to appropriate exercise programming. If, due to COVID-19 public health restrictions, community based programming cannot occur, the exercise sessions will be delivered online by fitness professionals.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of cancer
* are over the age of 18 years
* are able to participate in mild levels of activity
* are about to have treatment, are currently having treatment, or have had cancer treatment within the last 5 years
* can read/write in English
* can access online programs, if necessary, to participate in the exercise programs.

Exclusion Criteria:

* unable to read/write in English
* are unable to participate in exercise
* for online programs, do not have internet or computer access

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Minutes Per Week | Baseline to one-year
  Change in number of participants meeting Guidelines for Physical Activity of 150 minutes per week of moderate intensity exercise, based on accelerometer data from commercially-available activity tracker.

SECONDARY OUTCOMES:
Body Composition | Baseline to post 12-week exercise intervention
  Change in body mass index (BMI)
Aerobic Endurance | Baseline to post 12-week exercise intervention
  Change in 6-minute walk test (m) or 2 minute step test (steps) results
Upper extremity grip strength | Baseline to post 12-week exercise intervention
  Change in hand-grip dynamometry (kg)
Functional performance test | Baseline to post 12-week exercise intervention
  Change in sit-to-stand (number of repetitions in 30 seconds)
Upper extremity flexibility | Baseline to post 12-week exercise intervention
  Change in active shoulder flexion range of motion (degrees)
Lower extremity flexibility | Baseline to post 12-week exercise intervention
  Change in sit-and-reach test (cm)
Balance | Baseline to post 12-week exercise intervention
  Change in one legged stance test (seconds)
Symptom tracking | Baseline to one year
  Change in fatigue, mood, and QOL, recorded via m-Health app
Cancer related symptoms | Baseline to one year
  Change in Edmonton Symptom Assessment Scale.
  - scale is from 0-10, where 0 means the symptom is absent and 10 means the worst possible severity of the symptom is being experienced.
Subjective reporting of average weekly physical activity | Baseline to one year
  Change in Godin Leisure Time Exercise Questionnaire
General Health-related Quality of Life | Baseline to one year
  Change in EuroQual - 5Dimensions (EQ-5D) tool
  - first section is a questionniare; last section uses a scale from 0-100, where 0 means the worst health imaginable and 100 means the best health imaginable.
Fatigue | Baseline to one year
  Change in Functional Assessment of Chronic Illness Therapy - Fatigue subscale
  - scale is from 0-4, where 0 means "not at all" and 4 means "very much".
General well-being | Baseline to one year
  Change in Functional Assessment of Cancer Therapy - General subscale
  - scale is from 0-4, where 0 means "not at all" and 4 means "very much".
Cognition | Baseline to one year
  Change in Functional Assessment of Cancer Therapy - Cognitive subscale
  - scale is from 0-4, where 0 means "never" and 4 means "several times a day" (experiencing symptoms).
Barriers and facilitators to exercise participation | Baseline to one year
  Change in Exercise Barriers and Facilitators questionnaire
Exercise adherence | Baseline to one year
  Adherence to exercise programming (attendance at sessions)
Program implementation and evaluation | Baseline to one year
  RE-AIM: program reach, effectiveness, adoption, implementation and maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Culos-Reed, PhD, Principal Investigator — University of Calgary; Margaret L McNeely, PhD, Principal Investigator — University of Alberta; Melanie Keats, PhD, Principal Investigator — Dalhousie University
Locations (3):
- Canada (3):
  - Health and Wellness Lab, University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Dalhousie University, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No
No plan at this time to share IPD outside of the research team.

REFERENCES:
- [Derived] Culos-Reed N, Wagoner CW, Dreger J, McNeely ML, Keats M, Santa Mina D, Cuthbert C, Capozzi LC, Francis GJ, Chen G, Ester M, McLaughlin E, Eisele M, Sibley D, Langley J, Chiekwe J, Christensen T; EXCEL Project Team. Implementing an exercise oncology model to reach rural and remote individuals living with and beyond cancer: a hybrid effectiveness-implementation protocol for project EXCEL (EXercise for Cancer to Enhance Living Well). BMJ Open. 2022 Dec 29;12(12):e063953. doi: 10.1136/bmjopen-2022-063953. PMID 36581419